CLINICAL TRIAL: NCT00713622
Title: A Multicentre, Randomised, Active Comparator, Parallel Group Study To Compare The Effect On Cognition Of Adjunctive Therapy With Zonisamide Versus Sodium Valproate
Brief Title: Comparing The Effect On Cognition Of Adjunctive Therapy With Zonisamide Versus Sodium Valproate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-E044-406; 2007-005313-19 (EudraCT Number)
Record Dates: First submitted 2008-07-08; First posted 2008-07-11 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Partial; onset; seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Zonisamide; Valproic Acid; Epilim

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Zonisamide
- 2 (Active Comparator)
  Interventions: Drug: Sodium valproate

INTERVENTIONS:
Drug: Zonisamide — Capsules of 25mg, 50mg and 100mg zonisamide will be supplied. Dosing will be twice a day.
  Other Names: Zonegran
  Arms: 1
Drug: Sodium valproate — Crushable tablets of 100mg and enteric coated tablets of 200mg and 500mg will be supplied. Dosing will start at 600mg/day, increasing to the minimally effective dose, the maximum tolerated dose, or 2500mg/day, whichever is the lowest.
  Other Names: Epilim
  Arms: 2

SUMMARY:
Zonisamide (Zonegran) and sodium valproate (Epilim) are both medicines approved to treat epilepsy. The purpose of this study is to find out the extent to which zonisamide may affect memory and concentration, compared to sodium valproate.

DETAILED DESCRIPTION:
Zonisamide (Zonegran) and sodium valproate (Epilim) are both medicines approved to treat epilepsy.

The purpose of this study is to find out the extent to which zonisamide may affect memory and concentration, compared to sodium valproate. This will be investigated using cognitive tests which are performed on a computer screen. Either zonisamide or sodium valproate will be added as a second medicine to the one patients are currently taking, carbamazepine (Tegretol), which will be continued throughout the study.

It is planned that about 80 people across Europe will take part in this study. For the purpose of the study, patients will need to go to the study doctor's clinic 4 times and have 5 telephone calls. Involvement in the study might be as long as 20 weeks, but it could be as short as 12 weeks. The length of the study and number of visits will depend on whether patients have an accurate recording of previous seizures already, how many seizures they have during the study, and whether they decide to continue or to stop treatment after the study is completed.

Adult subjects with a clinical diagnosis of non-symptomatic (i.e., idiopathic or unknown cause) localisation-related epilepsy, with partial onset seizures with or without secondary generalisation, who are receiving fixed dose carbamazepine as their only therapy or can be transferred to carbamazepine (as their only therapy) in the two months before the study baseline. Subjects must require addition of another anti-epileptic drug (AED) to their anti-epileptic therapy, either because they continue to have seizures (i.e., are not controlled), or because they wish to switch to another AED for other reasons (e.g., they tolerate another drug better).

ELIGIBILITY:
Inclusion criteria:

1. Subjects with a clinical diagnosis of non-symptomatic (i.e., idiopathic or cryptogenic) localisation-related epilepsy with partial onset seizures with or without secondary generalisation according to International League Against Epilepsy (ILAE) classification27. Diagnosis should be clinically established by history, by previous electroencephalogram (EEG) and by previous magnetic resonance imaging or computer tomography of the brain, consistent with localisation related epilepsy. No lower or upper limit of baseline seizures is defined.
2. Able and willing to sign informed consent form (ICF) in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines.
3. Male or female subjects aged ≥18 years.
4. Subjects taking carbamazepine as monotherapy at baseline or who can be transferred to carbamazepine monotherapy in the two months before the Screening Visit. Dose of carbamazepine is within that recommended by the SPC. Carbamazepine dose has not been altered during the previous 2 weeks prior to the start of the Baseline Period, or 6 weeks if the Baseline Period is to be shortened due to the availability of a retrospective seizure history. The carbamazepine dose is to remain stable throughout the study.
5. Subjects requiring addition of another AED, either because they continue to have seizures (are refractory), or because they wish eventually to switch to another AED for other reasons after the study completion (e.g. tolerability reasons).
6. Female subjects of childbearing potential must not be pregnant (as confirmed by negative serum beta-human chorionic gonadotropin (βHCG) at screening and negative urine pregnancy test at baseline and during the study), must not be lactating and must use a medically acceptable form of contraception during the study and for at least 1 month after discontinuation of study drug. Medically acceptable contraception is defined here as:

   * High dose combined oral contraceptive (OC) pill (50µg of oestrogen preparation)
   * Documented surgical sterilisation or documented vasectomised sexual partner
   * Intrauterine device in place for at least 3 months and not exceeding the documented replacement date. (If the replacement date is not available, the device must not have been in situ for more than 5 years).
   * Women more than 2 years post-menopause
   * Abstinence Examples of contraception NOT acceptable include, but are not limited to:· Conventional dose of combined OC (< 50µg oestrogen)
   * Progesterone-only OC
   * Contraceptive implant
   * Contraceptive patch
   * Progesterone injection
   * Barrier contraception:

     * Condom
     * Diaphragm
     * Sponge

Exclusion criteria:

1. Previous treatment with valproate or zonisamide.
2. Use of an AED other than carbamazepine less than 6 weeks prior to randomisation, and other than carbamazepine, zonisamide or sodium valproate during the study.
3. Hypersensitivity to zonisamide or valproate or their respective excipients.
4. Predisposing condition potentially altering the absorption, distribution or elimination of zonisamide or valproate.
5. Sulphonamide allergy.
6. Subjects with diagnosed idiopathic/primary generalised epilepsy or with results of clinical investigations or EEG that suggest idiopathic/primary generalised epilepsy.
7. History of status epilepticus within 12 months of screening whilst complying with AED therapy.
8. History of cluster seizures.
9. History of non epileptic seizures.
10. Use of benzodiazepines during the Baseline Period or during randomised treatment.
11. Regular treatment with antihistamines.
12. Use of ketogenic diet.
13. Use of acetazolamide, triamterene, vitamin C (>2g/day), regular antacids or other medicines associated with nephrolithiasis less than one month prior to randomisation or during the study.
14. Subjects with a vagal nerve stimulator implanted, or due to be implanted within the expected duration of the study.
15. Subjects expected to undergo any surgery within the expected duration of the study.
16. History of renal calculi or renal insufficiency (above the upper normal limits of creatinine).
17. Active psychiatric disease.
18. History of suicide attempt within last 2 years.
19. History of drug or alcohol abuse within the last 2 years.
20. History of cerebrovascular disease/stroke or transient ischemic attacks; progressive neurological disease; focal central nervous system pathology or behavioural disturbances that may impair the subject's ability to complete the neuropsychological tests; or previous or current brain neoplasm.
21. Neoplastic disease within the last 5 years except non-metastatic and adequately treated cutaneous squamous cell carcinoma.
22. Diagnosis of human immunodeficiency virus (HIV) or Hepatitis B or C.
23. Other clinically significant organic disease.
24. Female subjects who are lactating, pregnant or intending to become pregnant.
25. Subjects with history of demonstrated non compliance with medication or an inability to maintain a seizure diary.
26. Subjects considered by the Investigator not to be within normal cognitive limits.
27. Participation in clinical study within 30 days of screening.
28. Clinically significant laboratory value abnormalities at baseline.
29. Weight <40kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in 28-day seizure frequency at Week 12; response rate at 12 weeks. | Change from baseline to Week 12 in the Computerised Visual Searching Task Reaction Time (CVST) from the Ferum Psyche (FePsy) cognitive battery, which measures central information processing speed conducted at visits 2, 5 and 8.

SECONDARY OUTCOMES:
Safety will be assessed by the incidence of AEs and serious adverse events (SAEs); incidence of withdrawal for treatment emergent adverse events (TEAEs); physical and neurological examinations. | Visits 1 and Visit 8; vital signs and weight conducted at Visits 1,2,5 and 8; clinical laboratory tests Visit 1 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Yeates, Study Director — Eisai Limited
Locations (2):
- Universitae Klinik fur Neurologiet, Innsbruck, Austria
- Kuopio University Hospital, Kuopio, Finland